CLINICAL TRIAL: NCT01140698
Title: Amino Acid Profile in the Fetus and the Neonate
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Leah Leibovitch, Shaba Medical Center
Other Study IDs: SHEBA-10-7895-LL-SMC
Record Dates: First submitted 2010-06-08; First posted 2010-06-09 (Estimated); Last update posted 2010-06-09 (Estimated); Status verified 2010-06

CONDITIONS: Cord Blood Amino Acid Profile; Fetal Amino Acid Profile in Different Gestational Ages; Infant Amino Acid Profile at Day 3 and Discharge

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Term and preterm newborn infants: 5 infants of each gestational age of 24-42 weeks
  Interventions: Other: Blood sample on Guthrie paper from cord blood, and day 3 of life and before discharge

INTERVENTIONS:
Other: Blood sample on Guthrie paper from cord blood, and day 3 of life and before discharge — Mass spectroscopy on the blood sample that are taken as routine for the national inborn errors survey

SUMMARY:
Up-to-date, the preterm newborn nutrition is based on human breast milk or it's imitations. However, the growth rate is known to be reduced compared to the fetal growth rate. In order to attempt a better growth rate of the preterm newborn infants it is important to evaluate the metabolic components of the fetal blood and try to find components that might influence its growth.

Little is known of the metabolic components of the fetal blood, including amino acid profile. The aim of the study is to evaluate amino acid profile in the fetus blood in different gestational ages and compare it to post natal period.

ELIGIBILITY:
Inclusion Criteria:

* All new-born infants 5 of each gestational age

Exclusion Criteria:

* none

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Term and preterm newborn infants
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2010-07

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba medical center, Ramat Gan, Israel